CLINICAL TRIAL: NCT07308717
Title: Gabapentin And Breast Surgery Decision Architecture Randomization Trial (GABS-DART) Protocol
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-183
Record Dates: First submitted 2025-12-17; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; unilateral mastectomy; bilateral mastectomy; 25-183; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Standard of care
- Intervention Arm (Experimental): The study intervention will consist of modification to the pre-operative order set to remove gabapentin.
  Interventions: Other: Modification to Pre-operative Order Set

INTERVENTIONS:
Other: Modification to Pre-operative Order Set — Modification to the pre-operative order set to remove gabapentin
  Arms: Intervention Arm

SUMMARY:
This study aims to assess whether gabapentin should be a standard component of peri-operative pain control in mastectomy patients at Memorial Sloan Kettering Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Undergoing ambulatory extended recover (AXR) mastectomy (bilateral or unilateral) at the Josie Robertson Surgical Center (JSRC)

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1896 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2027-12-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
Amount of postoperative morphine milligram equivalents/MMEs required after mastectomy | Up to 46 months
  Determine the effect of peri-operative gabapentin use on pain control in the PACU operationalized as the top quartile of postoperative morphine milligram equivalents/MMEs required in participants undergoing mastectomy

CONTACTS AND LOCATIONS:
Overall Officials: James Flory, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk-Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org